CLINICAL TRIAL: NCT06857578
Title: REDO- A Novel Surgical Revision Technique for Suboptimal Weight Loss or Recurrent Weight Gain After Roux-en-Y Gastric Bypass
Brief Title: Revision Surgery for Suboptimal Weight Loss or Recurrent Weight Gain After Roux-en-Y Gastric Bypass
Acronym: REDO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other)
Responsible Party: Principal Investigator, Torsten Olbers, Professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07210-01
Record Dates: First submitted 2025-02-18; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: revisional bariatric surgery; Roux-en-Y gastric bypass
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Efficacy and safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total revision of Roux-en-Y gastric bypass (Experimental): A complete revision of the previously performed Roux-en-Y gastric bypass
  Interventions: Procedure: Total revision of Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Total revision of Roux-en-Y gastric bypass — 1. The entire previous gastric bypass construction is released from any adhesions and all parts of the small intestine are measured and assessed.
  2. All or parts of the first part of the intestine that food reaches after the gastric pouch (so-called Roux) is resected. The reason is that parts of the intestine that are considered to be of poor quality (for example, affected by a lot of adhesions or abnormally dilated) are removed. This can be about 1.5 meters of intestine, which corresponds to 10-25% of the entire length of the small intestine.
     The gastric pouch will be small (<30 ml).
  3. A new gastric bypass construction is constructed where the intestine receiving food from the esophagus (Roux) will be 1 meter, and the small intestine part from the closed stomach at least 1.5 meters.
  The remaining length of the small intestine below the jejuno-jejunal anastomosis should be minimum 3 meters.

SUMMARY:
The majority of those who undergo gastric bypass surgery have a good/sufficient weight loss, averaging 25-30% after 10-20 years (Adams TD NEJM -18). In a subgroup analysis in LABS, 5% of RYGB patients had an unfavourable weight development with an average of only up to 10% weight loss 7 years after surgery (Courcoulas et al, JAMA Surg -18). These data are in good agreement with data in the Scandinavian quality registry SOReg where 5-10% an insufficient weight loss/weight recurrence 10 years after gastric bypass (SOReg annual report -20).

Insufficient weight loss/weight recurrence after gastric bypass can for the individual, in addition to the negative effects on quality of life, mean that comorbidities to obesity are insufficiently controlled or recur. This applies not least to weight-related problems, such as osteoarthritis in the lower extremities where joint replacement surgery can be prevented by too high a body weight.

In summary, one in ten patients who undergo bariatric surgery with the gastric bypass method will therefore have an insufficient effect of the procedure in the long term. The first-line treatment is a review of what can be done with diet and exercise, which, however, usually has a very limited effect. In recent years, the addition of medications has become an alternative, but the effect is variable and insufficiently studied over a longer period of time. These medications are also not included in the high-cost coverage.

The surgical method that has so far gained the most popularity in gastric bypass reoperation is the so-called "distal gastric bypass". In distal gastric bypass, the part of the intestine where much of the nutrient absorption occurs is so short that all nutrients (fat) are not fully absorbed. Although this method can be effective for weight loss, it often has significant side effects such as diarrhea and deficiencies of minerals and fat-soluble vitamins.

Over the past decade, knowledge about the mechanism of action of gastric bypass surgery has increased significantly. It is primarily changes in hunger and satiety signals from the gastrointestinal system to the brain that lead to sustained weight loss. Studies have shown that poorer weight loss is associated with a weaker response to satiety signals compared to those who lose more than average weight, where instead the response is strong.

Based on knowledge of the importance of satiety signals, initial experiences have been gained with a new type of revision surgery to amplify the effect in satiety signalling in gastric bypass patients with inadequate weight control. The results of these surgeries have generally been positive, even if not all achieved significant weight loss.

This project will systematically study whether a new type of revision surgery is safe and sufficiently effective to achieve the desired weight loss and improve comorbidity in patients who have responded inadequately or regained weight after gastric bypass surgery.

DETAILED DESCRIPTION:
This project aims to scientifically evaluate the risk/benefit ratio of a new type of reoperation/revision surgery for patient experiencing either a primarily poor response or late weight regain after Roux-en-Y gastric bypass surgery.

The scientific questions are:

Does the new surgical reconstruction lead to further weight loss? The primary endpoint for "successful" surgery is weight loss >10% of body weight 2 years after surgery.

What improvements in obesity comorbidities (e.g. type 2 diabetes, hypertension, dyslipidemia, sleep apnea, quality of life) can be achieved ?

Is the new surgical method associated with specific surgical risks and complications?

Is the new surgical method associated with an increased risk of nutritional deficiencies compared to primary gastric bypass?

Is the ability to eat and the bowel function affected in any way by the new surgical method?

An overall assessment will be made between investigators and the Data Safety and Monitoring Committee as to whether the positive effects of the procedure are sufficient in relation to the risks of the surgery.

Method:

We will conduct a case series with of 12 (6+6) gastric bypass patients with the new surgical method to achieve further weight loss and improved health.

Patients who have undergone gastric bypass surgery and have insufficient treatment effect (current weight <10% below the weight at the primary surgery) are identified at the outpatient clinic at the Department of Surgery, Vrinnevi Hospital in Norrköping. A clinically motivated investigation is carried out according to routine including a follow through X-ray to identify any anatomical defects in the gastric bypass construction or a gastro-gastric fistula.

If nothing abnormal emerges, it is further ensured that the patients have completed the usual intervention with lifestyle factors (diet and exercise) for optimized effect of the surgery. Patients will be informed that there are pharmacological treatments for weight loss (new drugs that are, however, not included in the high-cost coverage for this indication).

If, after the above, there is an agreement in the multidisciplinary team that revision surgery may be indicated and interest in treatment for the purpose of weight loss remains, the patients are asked about interest in participating in this study.

Patients will be thoroughly informed verbally during an outpatient visit and receive written research person information and plenty of time to ask questions. After a reasonable time for reflection and the opportunity to ask supplementary questions, an informed consent is signed if the attitude remains positive.

Basic investigation and supplementary study-specific information with validated questionnaires are obtained:

* Information about eating-related symptoms and so-called "dumping" with DSS (Dumping Severity Score)
* Information about gastrointestinal symptoms with GSRS (Gastrointestinal Symptom Rating Score)
* Blood samples in the quality registry SOReg are taken according to clinical routine as well as clinical information about, for example, current diseases and medication.

The usual preoperative preparation for the procedure then takes place, including at least 2 weeks of low calorie diet for preoperative weight loss. The keyhole surgical procedure includes:

1. The entire gastric bypass construction is exposed and released from any adhesions. All limbs of the small intestine are measured and assessed for quality.
2. All or parts of the first part of the intestine (the so-called Roux limb) is resected. The reason is that parts of the intestine may be of poor quality (for example, affected by adhesions or abnormally dilated) are removed. This can be about 1.5 meters of intestine, which corresponds to 10-25% of the entire length of the small intestine.

All or parts of the first part of the Roux-limb will be preserved if necessary to avoid having a too short total intestine length.

The gastric pouch should be small (<30 ml).

A new gastric bypass construction is constructed where the Roux limb is 1 meter long, and the small intestine section from the bypassed stomach is at least 1.5 meters long.

During the operation it is verified that the common limb (with full nutrient absorption) is at least 3 meters long to avoid malnutrition.

. The operation is performed under general anesthesia and the time for the operation itself is estimated to be between 90 and 120 minutes. After surgery, the patient is mobilized freely and is allowed to drink freely. Normally, the patient is discharged from the ward the day after the operation if everything has been uncomplicated. Sick leave is estimated to be between 2 and 3 weeks. Progress of the diet to regular solid food takes place over a month according to routine for primary gastric bypass surgery.

How does the project differ from standard care:

Usually health care is cautious about further surgical interventions in patients having regained weight after gastric bypass. However, revision surgeries such as "distal gastric bypass" or other surgical reconstructions have been performed in some clinics.

The surgical method to be studied in this project takes into account recently achieved knowledge about the mechanism of action of gastric bypass surgeries. By resecting the first part of the small intestine (1-1.5 meters) and performing a "new gastric bypass", this leads to:

1. The food becomes exposed to more distal small intestine. Distal exposure is associated with increased release of gastrointestinal hormones (including GLP-1 and PYY). These gastrointestinal hormones signal satiety acts via the hypothalamus, and this is a central mechanism of action in gastric bypass. Patients with poor weight loss after gastric bypass have been shown to have a weak response in this mechanism and those with good weight loss have strong signalling.
2. bile and gastric juices in the so-called "bilio-pancreatic limb" that connects the bypassed part of the stomach with the small intestine are lengthened. This has also been shown to be associated with increased release of gastrointestinal hormones (GLP-1, PYY) and greater weight loss. Bile and gastric juices in the intestine without concomitant food is a strong trigger for the release of satiety signals.
3. Any flaw in the primary gastric bypass construction that could contribute to an "incorrect" eating pattern (more sweet, fatty and liquid calories which is associated with weight gain) is corrected.
4. The absolute majority of the small intestine is preserved in the abdominal cavity and restoration of the anatomy is possible.

Previous experience with the intervention:

In a case series, conducted as a pilot project at Sahlgrenska University hospital in Gothenburg, Sweden the responsible researcher has operated on a dozen patients with total revision of the gastric bypass construction. Most often, it was a combined situation with suspected dysfunction of the gastric bypass and unsatisfactory weight effect. In those who were operated on with the new technique, the weight dropped on average from 127 to 101 kg (range for weight loss 2-54 kg) with varying follow-up times of up to several years. The patients' subjective assessment was: Two had unsatisfactory weight development (no or very limited weight loss, but no longer continued weight gain), The others were partially or completely satisfied with their weight development.

One patient had a lot of adhesions around the small intestine in connection with the revision surgery and developed adhesions again, which is why he ultimately needed surgery to restore normal anatomy after gastric bypass. Restoring normal anatomy is therefore still possible after this type of revision surgery, as at most 1-1.5 m of the length of the small intestine (normal length 6-11 m) is resected.

In none of the cases that underwent total revision did we note a tendency to nutritional deficiencies beyond what is seen after primary gastric bypass. No serious surgical complications arose in connection with the pilot series.

Data collection:

* weight, height, waist circumference, blood pressure
* inventory of comorbidities (e.g. medication for diabetes, high blood pressure, high blood lipids, sleep apnea, joint problems, inflammation).
* blood tests for comorbidities (fasting blood sugar, HbA1c, insulin, blood lipids, hs-CRP and blood status.
* blood sampling for vitamins and minerals.
* questionnaires for quality of life (standard for bariatric surgery)
* additional study-specific questionnaires for eating function and dumping (DSS) and gastrointestinal function (GSRS)

ELIGIBILITY:
Inclusion Criteria:

* Body weight within 10% of initial weight
* >2 year after primary Roux-en-Y gastric bypass procedure
* Able to comprehend intended benefits and risks
* Understand the Swedish language
* Not responding sufficiently to life style intervention
* Be aware about available pharmacological interventions

Exclusion criteria:

* Inflammatory bowel disease
* Below 25 or above 60 years of age

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2035-01-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss (kg) | 2 years
  We will consider the experimental procedure effective provided that 80% of participants lose at least 10% of preoperative weight

SECONDARY OUTCOMES:
Complication to surgery | 2 years
  Peri- or postoperative complications
Side effects to the gastro-intestinal reconstruction | 2 years
  Diarrhoea, malnutrition
Change in obesity comorbidity | 2 years
  Diabetes mellitus type 2, Hypertension, Hyperlipidemia, Obstructive Sleep Apnea, Joint pain
Waist circumference | 2 years
  In centimeter. Measured between lowest rib and iliac anterior/superior spina
Change in physical quality of life | 2 years
  RAND36 (Research AND Development). Four subscales measured from 0-100 where a higher score is better.
Change in mental quality of life | 2 years
  RAND36 (Research AND Development). Four subscales from 0-100 where a higher score is better.
Patient Reported Experience Measure | 2 years
  As measured in the Scandinavian Obesity Surgery Registry (SOReg)
Nutritional deficienies | 2 years
  Blood concentrations and proportion of participants having abnormal levels of Vitamin D, Ionized Calcium, Vitamin B12, Folate, Iron, Ferritin, Total Iron Binding Capacity, Albumin.

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Olbers, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Dept of Surgery, Vrinnevi hospital, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
Data protection legislation in Sweden